CLINICAL TRIAL: NCT02982811
Title: Intelligent Activity-based Client-centred Training
Acronym: i-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PXL University College (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); Ziekenhuis Oost-Limburg (Other); Hasselt University (Other)
Responsible Party: Principal Investigator, Els Knippenberg, Researcher and PhD student, PXL University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: i-ACT2
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Central Nervous System Diseases; Aged
Keywords: Activity-based; Client-centred; Rehabilitation; Quality of life
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Therapy as usual, i.e. occupational therapy, physiotherapy, etc.
- Experimental group (Experimental): Therapy as usual together with 3x45min training with i-ACT system during 6 weeks.
  Interventions: Device: i-ACT

INTERVENTIONS:
Device: i-ACT — 3x 45 min training with i-ACT system (analytical and functional training) during 6 weeks, additional to therapy as usual (i.e. occupational therapy, physiotherapy, etc.)
  Arms: Experimental group

SUMMARY:
The purpose of this study is to determine whether additional therapy with i-ACT system is effective in the training of functional skills in persons with central neurological diseases (e.g. multiple sclerosis, stroke, spinal cord injury, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of central nervous system disease (e.g. multiple sclerosis, stroke, spinal cord, etc.)
* Be able to understand and respond to questions in Dutch
* Actively involved in a rehabilitation programme in the participating rehabilitation centres
* Have a dysfunction in upper and/or lower limb and/or core stability
* Specifically for multiple sclerosis: min. of one month without corticosteroids
* Specifically for stroke and spinal cord: min. 3 months post injury

Exclusion Criteria:

* Severe spasticity which prevent performing basic functional exercises
* Severe cognitive and communicative impairment which prevent the person to understand and respond to Dutch instructions
* Severe visual impairment, e.g. blindness, cataract, etc.
* Pregnancy
* Persons who use an electrical wheelchair, who can not transfer safely into a normal chair and perform the exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of upper extremity
Short Form 36 (SF-36) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of general health status and quality of life

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) | After 6 weeks of training, only persons in experimental group
  Evaluation of motivation towards using the system in neurorehabilitation
Manual Ability Measure (MAM-36) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of performance of manual tasks
Modified Fatigue Impact Scale (MFIS) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of fatigue
Trunk Impairment Scale (TIS) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of sitting, standing and core stability
Active Range of Motion (AROM) | At baseline, after 3 and 6 weeks of training, and 6 weeks follow-up
  Evaluation of active range of motion
Canadian Occupational Performance Measure (COPM) | At baseline, after 6 weeks of training, and 6 weeks follow-up
  Evaluation of self-perception of performance of ADL tasks

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Spooren, Prof. Dr., Study Director — Centre of Expertise - Innovation in Care
Locations (4):
- Belgium (4):
  - Jessa Hospital - rehabilitation campus St-Ursula, Herk-de-Stad, Limburg
  - Ziekenhuis Oost Limburg, Lanaken, Limburg
  - Revalidatie en MS centrum, Overpelt, Limburg
  - St-Trudo hospital, Sint-Truiden, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knippenberg E, Timmermans A, Coolen J, Neven K, Hallet P, Lemmens J, Spooren A. Efficacy of a technology-based client-centred training system in neurological rehabilitation: a randomised controlled trial. J Neuroeng Rehabil. 2021 Dec 28;18(1):184. doi: 10.1186/s12984-021-00977-2. PMID 34961531